CLINICAL TRIAL: NCT00764556
Title: Phase II Study of Safety and Feasibility of Intensive Blood Glucose Control With Insulin on Acute Medical Wards
Acronym: IPS2008
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Dr Emma Baker, St George's, University of London
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGH-ClinPharm-1; EudraCT 2007-004956-35; Ethics 07/H0715/93
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: COPD; Hyperglycemia
Keywords: Glucose; Insulin; COPD; Exacerbations; Tight glycaemic control; Acute hospital ward
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hyperglycemia; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tight glycaemic control (Experimental): Intravenous or subcutaneous insulin to control blood glucose to 4.4-6.5mM
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Intravenous insulin (actrapid) Subcutaneous insulin (aspart, glargine, detemir)

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) are commonly admitted to hospital with exacerbations of their lung disease. A combination of the acute illness and treatment with oral steroids causes a rise in blood sugar. Patients with high blood sugar do worse than those with normal blood sugar. The aim of this study is to develop a safe and effective protocol for tight control of blood glucose with insulin on acute medical wards outside the intensive care environment. This will allow us to perform a formal trial to determine whether blood glucose control with insulin reduces death and complications from COPD exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of AECOPD as primary cause for admission
* Able to enter study within 24 hours of admission

Exclusion Criteria:

* Intensive care unit admission
* Moribund or not for active treatment
* Admission expected to last <48 hours
* Unable or unwilling to give informed consent
* Known Type I diabetes mellitus
* Patients with reduced awareness of hypoglycaemia including reduced Glasgow coma scale or those taking beta blockers
* Patients with renal or hepatic failure at increased risk of hypoglycaemia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The frequency of severe hypoglycaemia - Neuroglycopenic symptoms (other than mild agitation) responsive to administration of carbohydrate | During trial

SECONDARY OUTCOMES:
The frequency of symptomatic hypoglycaemia (capillary glucose≤3.3mM AND symptoms consistent with hypoglycaemia) | During trial
The frequency of asymptomatic hypoglycaemia (capillary glucose≤3.3mM without any symptoms consistent with hypoglycaemia). | During treatment
Mean 24 hour capillary glucose concentrations | During treatment
Proportion of capillary glucose measurements in target range (4.4-6.5mM) | During treatment
Comparison of capillary blood glucose measurements to those obtained from the Guardian REAL®-time continuous glucose monitoring system | During monitoring
Comparison of rates of detection of hypoglycaemia by capillary and continuous blood glucose monitoring | During monitoring
Quantification of acceptability of the study intervention to patients | during study

CONTACTS AND LOCATIONS:
Overall Officials: Emma H Baker, PhD, FRCP, Principal Investigator — St George's, University of London
Locations (1):
- St George's Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Baker EH, Janaway CH, Philips BJ, Brennan AL, Baines DL, Wood DM, Jones PW. Hyperglycaemia is associated with poor outcomes in patients admitted to hospital with acute exacerbations of chronic obstructive pulmonary disease. Thorax. 2006 Apr;61(4):284-9. doi: 10.1136/thx.2005.051029. Epub 2006 Jan 31. PMID 16449265
- [Derived] Archer JR, Misra S, Simmgen M, Jones PW, Baker EH. Phase II study of tight glycaemic control in COPD patients with exacerbations admitted to the acute medical unit. BMJ Open. 2011 Jul 23;1(1):e000210. doi: 10.1136/bmjopen-2011-000210. PMID 22021788